CLINICAL TRIAL: NCT07292597
Title: How Do Individual Differences in Circadian Rhythms Influence Time Perception?
Brief Title: Circadian Timing and Time Perception in Healthy Adults
Acronym: ChronoTime
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1-10-72-108-25; 10.46540/4256-00108B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2025-11-14; First posted 2025-12-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Circadian Rhythm; Time Perception
Keywords: chronotype; circadian misalignment; duration discrimination; time production; time estimation

STUDY DESIGN:
Intervention Model Description: Two-period, two-sequence (AB/BA) crossover. Each participant completes both sessions: circadian-congruent timing and circadian-incongruent timing. Session order is randomized; sessions occur morning and evening on the same day with a substantial interval and standardized pre-session restrictions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB - Congruent → Incongruent (Experimental): rossover sequence AB. Participants first complete a circadian-congruent session (morning types in the morning; evening types in the evening), followed by a circadian-incongruent session (opposite time). Intervention administered: Behavioral - Session timing relative to chronotype.
  Interventions: Behavioral: Session timing relative to chronotype
- Sequence BA - Incongruent → Congruent (Experimental): Crossover sequence BA. Participants first complete a circadian-incongruent session (opposite of their preferred time), then a circadian-congruent session. Intervention administered: Behavioral - Session timing relative to chronotype.
  Interventions: Behavioral: Session timing relative to chronotype

INTERVENTIONS:
Behavioral: Session timing relative to chronotype — Two-period, two-sequence crossover manipulation of testing time. Each participant completes both sessions: (1) circadian-congruent timing (morning types tested in the morning; evening types in the evening) and (2) circadian-incongruent timing (opposite time). Session order is randomized (AB/BA). Sessions are run morning and evening on the same day with a substantial interval; no visible clocks; 12-h pre-session caffeine/strenuous-exercise restriction; standardized lab light/temperature. Primary outcomes: time-estimation/production bias and PVT lapses/RT.
  Other Names: Circadian alignment; Circadian misalignment; Timing condition

SUMMARY:
This study examines how a person's natural daily rhythm ("chronotype") affects the way time is experienced and judged. Healthy Danish-speaking adults (23-45 years) who are clearly morning-type or evening-type will complete two lab sessions in a crossover design: one at their preferred time of day (e.g., morning for morning-types) and one at the opposite time (misaligned). In each session, participants do brief computerized tasks that measure time estimation/production, vigilance (psychomotor vigilance task), decision-making, and responses to social information, plus simple color-vision tasks. Short questionnaires about sleepiness, mood, fatigue, and the subjective "passage of time" are collected before, during, and after testing. A subset will wear a wrist actigraphy device for one week beforehand to characterize sleep-wake patterns.

Testing is conducted under standardized lab conditions with scheduled breaks. The main goal is to determine whether time judgments and vigilance are less accurate during the misaligned session and whether decision-making and social responses also vary with circadian timing. Risks are minimal and mainly relate to temporary tiredness when tested at a non-preferred time; participants may stop at any time. Participation is voluntary. Data are pseudonymized and handled under GDPR. Participants receive DKK 300 after completing both sessions (pro-rated if they withdraw early). Results will be published regardless of outcome, and de-identified data/code will be shared after publication.This study examines how a person's natural daily rhythm ("chronotype") affects the way time is experienced and judged. Healthy Danish-speaking adults (23-45 years) who are clearly morning-type or evening-type will complete two lab sessions in a crossover design: one at their preferred time of day (e.g., morning for morning-types) and one at the opposite time (misaligned). In each session, participants do brief computerized tasks that measure time estimation/production, vigilance (psychomotor vigilance task), decision-making, and responses to social information, plus simple color-vision tasks. Short questionnaires about sleepiness, mood, fatigue, and the subjective "passage of time" are collected before, during, and after testing. A subset will wear a wrist actigraphy device for one week beforehand to characterize sleep-wake patterns.

Testing is conducted under standardized lab conditions with scheduled breaks. The main goal is to determine whether time judgments and vigilance are less accurate during the misaligned session and whether decision-making and social responses also vary with circadian timing. Risks are minimal and mainly relate to temporary tiredness when tested at a non-preferred time; participants may stop at any time. Participation is voluntary. Data are pseudonymized and handled under GDPR. Participants receive DKK 300 after completing both sessions (pro-rated if they withdraw early). Results will be published regardless of outcome, and de-identified data/code will be shared after publication.

DETAILED DESCRIPTION:
Background/Rationale. Circadian rhythms vary across individuals (chronotypes) and can be misaligned with social schedules. Both circadian timing and time perception influence cognition and behavior, yet within-person effects of circadian alignment on temporal judgments and related functions are not well characterized.

Objectives/Hypotheses. Primary: test whether circadian misalignment (testing at a non-preferred time) increases time-estimation/production bias and reduces vigilance versus aligned testing. Secondary: assess effects on temporal variability, duration discrimination, decision-making strategies, social conformity, and simple color-perception measures (white-point/unique-hue).

Design. Randomized, two-condition crossover trial with within-subject comparison of circadian-congruent vs incongruent sessions (order counterbalanced). Sessions occur on the same day (morning and evening) with a substantial break; no visible clocks; caffeine/exercise restrictions prior to testing. A subset (n≈60) completes 7-day actigraphy and sleep diary.

Participants. Healthy adults, 23-45 years, Danish-speaking, clear morning or evening chronotype (MEQ/MCTQ). Key exclusions: shift work, recent trans-meridian travel, sleep/neurologic/psychiatric disorders, medications affecting sleep/cognition, intermediate chronotype.

Intervention. Behavioral manipulation of testing time relative to chronotype (congruent vs incongruent) in a crossover design.

Outcomes.

Primary: (1) Time-estimation/production bias across 10-60 s targets; (2) Psychomotor vigilance task (lapses, RT).

Secondary: Time-estimation variability (CV), duration discrimination threshold, passage-of-time ratings, KSS sleepiness, mood/fatigue scales, information-conformity effect, decision-making metrics, color-perception indices (white-point/unique-hue).

Outcome time frame: per session; within-subject contrast (incongruent-congruent).

Sample size/Analysis. Target N≈128. Within-subject models test condition effects, with chronotype and session order as factors; missing data handled with mixed-effects models. Alpha=0.05 (two-sided).

Data management/Sharing. Pseudonymized data stored per AU policy/GDPR. De-identified datasets and analysis code will be shared in an open repository within 12 months of primary publication.

Risk/Benefit. Minimal risk (temporary tiredness). Potential benefits include improved understanding of circadian influences on cognition with implications for scheduling and performance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 23 to 45 years
* Able to understand and communicate in Danish
* Completed at least upper secondary education (e.g., gymnasium)
* Categorized as either a Morning Type (MT) or Evening Type (ET) based on standardized chronotype assessments:

  * Munich Chronotype Questionnaire (MCTQ):

    * MT: sleep midpoint on free days (MSFsc) ≤ 03:00
    * ET: sleep midpoint on free days (MSFsc) ≥ 05:00
  * Morningness-Eveningness Questionnaire (MEQ):

    * One of four defined chronotype categories (definitely morning, moderately morning, moderately evening, definitely evening).

Exclusion Criteria:

* Current engagement in shift work, rotating schedules, or other forms of irregular sleep-wake timing
* Diagnosis of any neurological, psychiatric, or sleep-related disorder (e.g., insomnia, narcolepsy, sleep apnea)
* Use of medications that affect sleep, alertness, or circadian functioning (e.g., melatonin, stimulants, antidepressants)
* International travel across time zones within the four weeks preceding study participation
* Are classified as having an intermediate chronotype based on validated chronotype assessments (MCTQ or MEQ), as this group does not provide the necessary contrast to evaluate circadian alignment effects.

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 128 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Time estimation bias | Day 1 (once during each of the two laboratory sessions: morning and evening)
  Signed percent error across 10, 30, and 60 s trials with a fixation cross: ((estimated - target)/target) × 100. Three trials per duration; session-level mean computed. Primary contrast: incongruent - congruent (within-subject). Higher values = overestimation.

SECONDARY OUTCOMES:
Psychomotor Vigilance Task (PVT) lapses (count) | Day 1 (once during each of the two laboratory sessions: morning and evening)
  Number of lapses (reaction time > 500 ms) during a 10-minute PVT. Session-level count. Primary contrast: incongruent - congruent (within-subject). Secondary PVT metrics (median RT, 10% slowest RT) analyzed separately.
Time production bias (neutral stimuli, 10-60 s) | Day 1 (once during each of the two laboratory sessions: morning and evening)
  Signed percent error for produced intervals vs targets (10, 30, 60 s). Three trials per duration; session-level mean. Contrast: incongruent - congruent (within-subject).
Duration discrimination threshold (2AFC adaptive) | Day 1 (once during each of the two laboratory sessions: morning and evening)
  JND (ms or % of standard) from a 2-interval, 3-down/1-up staircase with sub-second to few-second standards; session-level threshold. Contrast: incongruent - congruent.
Subjective passage-of-time rating (VAS 0-100) | Day 1 (pre-, mid-, and post-session ratings during each of the two laboratory sessions)
  VAS rating of "how fast time felt" collected pre/mid/post session; session-level mean or change from baseline. Contrast: incongruent - congruent.
Decision-making exploration rate (%) - Alien Game | Day 1 (once during each of the two laboratory sessions: morning and evening)
  Percent exploratory choices and total reward in a computerized multi-armed task; session-level metrics. Contrast: incongruent - congruent.
Social conformity effect (% shifts toward majority) | Day 1 (once during each of the two laboratory sessions: morning and evening)
  Proportion of responses shifted toward displayed majority opinion vs own baseline on perceptual judgments; session-level effect size. Contrast: incongruent - congruent.

CONTACTS AND LOCATIONS:
Locations (1):
- Cognition and Behavior Lab, Aarhus, Denmark